CLINICAL TRIAL: NCT04574336
Title: Scandinavian Humeral diAphyseal Fracture Trial - A Pragmatic Randomized Controlled Trial
Brief Title: Scandinavian Humeral Diaphyseal Fracture Trial
Acronym: SHAFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Zealand University Hospital (Other); Oslo University Hospital (Other); Helse Stavanger HF (Other Government); Sahlgrenska University Hospital (Other); Uppsala University Hospital (Other); Odense University Hospital (Other); Hospital of Southern Jutland (Other); Slagelse Hospital (Other); Aalborg University Hospital (Other); University Hospital, Umeå (Other); Nordsjaellands Hospital (Other); Holbaek Sygehus (Other); Aarhus University Hospital (Other); Copenhagen University Hospital at Herlev (Other); University Hospital Bispebjerg and Frederiksberg (Other); Viborg Regional Hospital (Other); Karolinska University Hospital (Other); Danderyd Hospital (Other); Tampere University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHAFT
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-06

CONDITIONS: Fracture Humerus of Shaft
Keywords: Humeral shaft fracture; Diaphysis; Fracture fixation; Fracture Healing; Aged; Randomized Controlled Trial; Comparative study
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Treatment (Experimental): Primary surgery of humeral shaft fracture with surgeons choice of osteosynthesis method
  Interventions: Procedure: Surgical treatment
- Non-surgical treatment (Active Comparator): Treatment of humeral shaft fracture with sling and/or functional brace
  Interventions: Device: Non-surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — We anticipate that surgical treatment will include plate osteosynthesis (MIPO and ORIF), intramedullary nailing (antegrade and retrograde) and external fixation. Plate and nail types, screw configuration and surgical approaches will be decided by the surgeon. The procedure will be conducted or supervised by a senior consultant.
  Arms: Surgical Treatment
Device: Non-surgical treatment — Non-surgical treatment will include sugar tong, splint, plaster splints, hanging casts, or functional bracing as the Sarmiento brace and will be worn until a surgeon removes it. If the surgeon deems it appropriate, participants will be offered to undergo early secondary surgery with a surgical procedure of their choice. The participants will be recorded and the reason will be noted. We anticipate the surgical procedures will be similar to the previous mentioned and perhaps with the addition of bone graft.
  Arms: Non-surgical treatment

SUMMARY:
This pragmatic multicenter randomized controlled trial (RCT) includes adult participants with an acute humeral shaft fracture to compare surgical fixation of humeral shaft fracture to non-surgical treatment with early identification and treatment of delayed union by a patient-reported outcome after 52 weeks. The trial population of 287 participants The trial population is divided in two age-groups due to the changes in DASH score by age. The definition of delayed union differs in the young and elderly population to consider dissimilarity in bone healing rates and the timepoint for crossover is therefor different between the groups. Participants will be randomized 1:1 between non-surgical treatment and surgical treatment. The primary outcome is the Disability of Arm, Shoulder and Hand (DASH) score at 52 weeks, and is assessor blinded. The secondary outcomes are DASH score earlier than 52 weeks, EQ-5D-5L, pain assessed by visual analogue score, Constant-Murley score including elbow range of motion and anchor-questions collected at all timepoints throughout the trial. All complications will be reported including; infection, nerve or vascular injury, surgical revisions (implant malpositioning, hardware failure, aseptic loosening and peri-implant fracture), major adverse cardiovascular events, other major adverse events and mortality. SHAFT will provide information on the effectiveness of two standard treatments for humeral shaft fractures, while taking the dilemmas within the population into account.

DETAILED DESCRIPTION:
We will conduct a pragmatic multicenter, randomized, controlled, outcome assessor-blinded, clinical superiority trial. The objective is to compare surgical fixation of humeral shaft fracture to non-surgical treatment with early identification and treatment of delayed union by a patient-reported outcome after 52 weeks. .

Null-hypothesis:

The DASH score at 52 weeks after surgical treatment is not superior to non-surgical treatment with the option of early crossover surgery in patients with humeral shaft fractures

The trial population is divided in two age-groups due to the changes in DASH score by age. The definition of delayed union differs in the young and elderly population to consider dissimilarity in bone healing rates:

1. SHAFT-Y for the young with an age cut-off of 18 to 64 years. The early identification and treatment of delayed union is set to 6 to 12 weeks
2. SHAFT-E for the elder with an age cut-off +65 years. The early identification and treatment of delayed union is set to 12 to 26 weeks

Sites from Denmark, Sweden and Norway have been recruited and spans from academic level I to level III trauma centers

287 patients (n=163 for SHAFT-Y, n=124 for SHAFT-E) with a humeral shaft fracture will be equally randomized to surgical treatment or non-surgical treatment in each group.

Patients admitted to the emergency department in one of the trial sites and fulfil the eligibility criteria, will be invited to enroll into the trial. They will be given time to consider and be scheduled for a consultation with a trial worker within 10 days. If written consent is obtained at the consultation, randomization will occur immediately after.

Treatment will be performed within 14 days after injury

* Surgical treatment. The specific treatment is decided by the treating surgeon/department
* Non-surgical treatment with the option of early secondary surgery from 6-12 weeks for SHAFT-Y and 12-26 weeks for SHAFT-E

Patients can be offered to undergo early crossover fixation with a surgical procedure of the surgeon's choice, if one of these criteria are met:

* Unacceptable pain experienced by the patient
* Severe pain with gross instability of the fracture site assessed by:
* Unable to en bloc elevate the arm due to clear fracture instability
* Gentle manipulation of the fracture site. Gentle manipulation should respect the risk of callus breakage
* Severe problems tolerating the brace, e.g. discomfort, skin irritation, wounds, hygiene problems.

The patients that undergo early crossover surgery will have the reason for crossover thoroughly noted. We anticipate the surgical procedures will be similar to the ones previously mentioned with the possible addition of bone graft.

A computerized database software, Research Electronic Data Capture (REDCap) will be used to generate an irreversible random allocation sequence and perform block randomization with selected block sized of 2 and 4, which will be stratified on site and age (18-64 and +65). Patients will be assigned to the trial with an allocation of 1:1 to either surgical treatment or non-surgical treatment. The trial worker acquires the allocated treatment from the central coordinator with randomization rights to REDCap. The trial worker then initiates the treatment, either by scheduling the surgery date or applying the chosen non-surgical method.

The two groups (SHAFT-Y and SHAFT-E) require individual sample size calculations. Two standard deviations (SDs) were obtained from the data of the FISH trial(13) and were separated in age groups of 18-64 years and 65 years and above. By the distribution-based approach, one half a SD corresponds to the minimal important change (MIC). The calculations are powered to detect a MIC of 7 points in the young and 10 points in the elderly group in DASH, respectively. Two independent means sample size calculation were performed. For SHAFT-Y the following data were included: Mean difference= 7.0, SD= 14.91, α= 0.05 and power= 0.8. For SHAFT-E the following data were included: Mean difference= 10.0, SD= 18.59, α= 0.05 and power= 0.8. Based on the preceding assumptions and including an attrition of 15%, the total sample size is estimated to 163 patients for SHAFT-Y and 124 patients for SHAFT-E.

Primary analysis Descriptive statistics will be used to report demographic data. Demographic data and outcome measures will be tested visually and statistically (i.e. Shapiro Wilks test). Numeric variables will be summarized by means, standard deviations and 95% confidence intervals (95% CI). Median and interquartile ranges will be used when normal distribution is not met. Categorical variables will be summarized by frequency and proportion. For group comparison with numerical data, a student's t-test will be used if data is normally distributed, otherwise a non-parametric test will be used. For categorical data a Chi-square test will be used for group comparison. An intention-to-treat (ITT) analysis of the primary outcome will be conducted by univariable linear regression, including all patients that do not meet the withdrawal criteria and will be conducted to minimize bias within results. A sensitivity analysis will test the effects of non-adherence to protocol by conducting a per-protocol analysis and includes only patients who comply with the protocol. For missing data points in an outcome measure, a multiple imputation analysis using predictive covariates (age, sex, smoking, alcohol, UCLA activity, ASA grade)(50-52) will be conducted to deal with nonresponse bias. For comparison we will carry out a sensitivity analysis excluding all the missing values.

Data will be considered statistically significant if p-values < 0.0471.

Secondary analysis In order to validate data a linear regression analysis will be computed with DASH score as the dependent variable and treatment modality as the independent variable. Additional regression analysis will be carried out between the early crossover group and the primary treatments. A multivariate regression analysis will be conducted to adjust for potential confounders. Variables adjusted for are: age, sex, smoking, alcohol, UCLA activity, ASA grade. Furthermore, we will analyze the longitudinal observations by applying a linear mixed effects regression model, including modality and time as well as a modality-time interaction as fixed effects and a random intercept for each patient. Data will be summarized as coefficients with 95% CIs and variance will be summarized as r-squares, adjusted r-squares, predicted r-squares, standard errors. Coefficients will be considered statistically significant if p-values < 0.05.

Outcome timepoints Subjective and objective outcome measures will be obtained at following time points: pre-injury, baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks, 2 years and 5 years.

ELIGIBILITY:
1. Fracture types 12A-C (OTA/AO classification)

   a. Includes minimal displaced extra-articular fracture extensions to the proximal humerus (less than a 1 cm or 45 degree angulation)
2. Treatment within 14 days from trauma
3. Age 18-64 years for SHAFT-Y and ≥65 years for SHAFT-E
4. Patients must understand the information given and be able to read and speak Danish, Swedish or Norwegian to complete the study paperwork

All fracture extensions involving the distal humerus and displaced fracture extensions involving the proximal humerus will not be included. Isolated fractures to the proximal or the distal end of the humerus are not eligible for screening. The proximal and distal end segments of the humerus are defined by squares of which the sides are the widest length of the epiphysis/metaphysis in question on the anterior-posterior view.

Exclusion criteria

1. Inability to give informed consent
2. Undisplaced shaft fracture (less than a cortex-wide displacement in all radiographic plane)
3. Vascular injury in ipsilateral arm
4. Polytrauma (defined as a trauma with one or more concurrent fractures to the upper extremities or other trauma absolute indications for surgical intervention)
5. Pathological fracture
6. Open fracture
7. BMI > 40
8. Health conditions preventing either treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 52 weeks
  A patient-reported outcome measure specific for physical function and symptoms of the upper limb (Disability of Arm, Shoulder and Hand-DASH). Scores range from 0 (no disability) to 100 (most severe disability)

SECONDARY OUTCOMES:
EuroQol-5 Domain (EQ-5D-5L) | Pre-Injury, 6 weeks, 12 weeks, 26 weeks, 52 weeks
  EuroQol questionnaire for patient reported outcome concerning health related quality of life measure. The score includes five dimensions with 5 levels from 1 (indicating no problem) to 5 (indicating extreme problem). EQ-5D-5L describes 3125 potential health states. A score of 11111 indicates having no problems in any of the dimensions and a score of 55555 indicates having extreme problems in all of the dimensions.
Rate of complications | Up to 52 weeks
  Complications after treatment will be recorded and include local complications, early general complication and mortality:
  * Local complications: Infection (needing antibiotic treatment with or without debridement), nerve or vascular injury, surgical revision (due to implant malpositioning, hardware failure, aseptic loosening or peri-implant fracture) and tolerance problems with brace (discomfort resulting in non-compliance of wearing the brace
  * Early general complications needing hospitalization within 12 weeks:
  Major adverse cardiac events (MACE) including myocardial infarction, heart failure, thromboembolism, cardiomyopathy and cardiac arrythmias.
  Other major adverse events including pneumonia, renal failure, electrolyte abnormality and deficiency anemia and other unforeseen reasons for hospitalization.
  • Mortality
Visual Analogue Scale (VAS) | Baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Visual analog scale is a pain score. Scores range from 0 (no pain) to 100 (worst pain).
Anchor question | 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Anchor questions will include Clinical anchor questions (CAQ), Retrospective Global Transition questions (RGTQ) and Binary Repeat Treatment (BRT).
  RGTQ and BRT will only be obtained at 52 weeks.
Constant-Murley score | 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Functional outcome with a 100-points scale. The higher the score, the higher the quality of the function.
Elbow range of motion | 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Range of motion is measured with a inclinometer.
Disabilities of the Arm, Shoulder and Hand (DASH) score | Pre-injury, 6 weeks, 12 weeks, 26 weeks
  A patient-reported outcome measure specific for physical function and symptoms of the upper limb (Disability of Arm, Shoulder and Hand-DASH). Scores range from 0 (no disability) to 100 (most severe disability)

OTHER OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 2 years, 5 years
  A patient-reported outcome measure specific for physical function and symptoms of the upper limb (Disability of Arm, Shoulder and Hand-DASH). Scores range from 0 (no disability) to 100 (most severe disability)
EuroQol-5 Domain (EQ-5D-5L) | 2 years, 5 years
  EuroQol questionnaire for patient reported outcome concerning health related quality of life measure. The score includes five dimensions with 5 levels from 1 (indicating no problem) to 5 (indicating extreme problem). EQ-5D-5L describes 3125 potential health states. A score of 11111 indicates having no problems in any of the dimensions and a score of 55555 indicates having extreme problems in all of the dimensions.
Radiological measurements | Baseline, 6 weeks, 12 weeks, 26 weeks, 52 weeks
  Radiographic images of the humeral shaft fracture will be assessed for fracture displacement, angulation, pattern, location and progression of radiological union.
Fracture instability | 6 weeks, 12 weeks
  Clinical sign of gross instability of the fracture site
Nonunion | Up to 52 weeks
  Gross mobility from the fracture site
Return to work | Up to 52 weeks
  Return to work is reported as a rate, from date of randomization until the date of first documented return to partial and full work.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarke Viberg, MD, PhD, Study Chair — Hospital Lillebaelt
Locations (22):
- Denmark (14):
  - Aabenraa Hospital, Aabenraa
  - Aarhus Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Aalborg-Farsø Hospital, Farsø
  - Herlev-Gentofte Hospital, Gentofte Municipality
  - New North Zealand Hospital, Hillerød
  - Holbæk Hospital, Holbæk
  - Kolding Hospital, Kolding
  - Zealand University, Køge
  - Odense Hospital, Odense
  - Slagelse Hospital, Slagelse
  - Viborg Regional Hospital, Viborg
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Norway (2):
  - Oslo University Hospital (Ullevål), Oslo
  - Stanvanger University Hospital, Stavanger
- Sweden (4):
  - Danderyd University Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Background] Kim SH, Szabo RM, Marder RA. Epidemiology of humerus fractures in the United States: nationwide emergency department sample, 2008. Arthritis Care Res (Hoboken). 2012 Mar;64(3):407-14. doi: 10.1002/acr.21563. PMID 22162357
- [Background] Ekholm R, Adami J, Tidermark J, Hansson K, Tornkvist H, Ponzer S. Fractures of the shaft of the humerus. An epidemiological study of 401 fractures. J Bone Joint Surg Br. 2006 Nov;88(11):1469-73. doi: 10.1302/0301-620X.88B11.17634. PMID 17075092
- [Background] Gosler MW, Testroote M, Morrenhof JW, Janzing HM. Surgical versus non-surgical interventions for treating humeral shaft fractures in adults. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008832. doi: 10.1002/14651858.CD008832.pub2. PMID 22258990
- [Background] Harkin FE, Large RJ. Humeral shaft fractures: union outcomes in a large cohort. J Shoulder Elbow Surg. 2017 Nov;26(11):1881-1888. doi: 10.1016/j.jse.2017.07.001. PMID 29054684
- [Background] Matsunaga FT, Tamaoki MJ, Matsumoto MH, Netto NA, Faloppa F, Belloti JC. Minimally Invasive Osteosynthesis with a Bridge Plate Versus a Functional Brace for Humeral Shaft Fractures: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Apr 5;99(7):583-592. doi: 10.2106/JBJS.16.00628. PMID 28375891
- [Background] van Middendorp JJ, Kazacsay F, Lichtenhahn P, Renner N, Babst R, Melcher G. Outcomes following operative and non-operative management of humeral midshaft fractures: a prospective, observational cohort study of 47 patients. Eur J Trauma Emerg Surg. 2011 Jun;37(3):287-96. doi: 10.1007/s00068-011-0099-0. Epub 2011 Apr 1. PMID 21837261
- [Background] Gottschalk MB, Carpenter W, Hiza E, Reisman W, Roberson J. Humeral Shaft Fracture Fixation: Incidence Rates and Complications as Reported by American Board of Orthopaedic Surgery Part II Candidates. J Bone Joint Surg Am. 2016 Sep 7;98(17):e71. doi: 10.2106/JBJS.15.01049. PMID 27605696
- [Background] Ramo L, Sumrein BO, Lepola V, Lahdeoja T, Ranstam J, Paavola M, Jarvinen T, Taimela S; FISH Investigators. Effect of Surgery vs Functional Bracing on Functional Outcome Among Patients With Closed Displaced Humeral Shaft Fractures: The FISH Randomized Clinical Trial. JAMA. 2020 May 12;323(18):1792-1801. doi: 10.1001/jama.2020.3182. PMID 32396179
- [Background] Hosseini Khameneh SM, Abbasian M, Abrishamkarzadeh H, Bagheri S, Abdollahimajd F, Safdari F, Rahimi-Dehgolan S. Humeral shaft fracture: a randomized controlled trial of nonoperative versus operative management (plate fixation). Orthop Res Rev. 2019 Sep 23;11:141-147. doi: 10.2147/ORR.S212998. eCollection 2019. PMID 31576178
- [Background] Oliver WM, Carter TH, Graham C, White TO, Clement ND, Duckworth AD, Molyneux SG. A prospective randomised controlled trial of operative versus non-operative management of fractures of the humeral diaphysis: the HUmeral Shaft Fracture FIXation (HU-FIX) Study protocol. Trials. 2019 Aug 5;20(1):475. doi: 10.1186/s13063-019-3576-0. PMID 31383027
- [Background] Kurup H, Hossain M, Andrew JG. Dynamic compression plating versus locked intramedullary nailing for humeral shaft fractures in adults. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD005959. doi: 10.1002/14651858.CD005959.pub2. PMID 21678350
- [Background] Driesman AS, Fisher N, Karia R, Konda S, Egol KA. Fracture Site Mobility at 6 Weeks After Humeral Shaft Fracture Predicts Nonunion Without Surgery. J Orthop Trauma. 2017 Dec;31(12):657-662. doi: 10.1097/BOT.0000000000000960. PMID 28708781
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Kunutsor SK, Barrett MC, Whitehouse MR, Blom AW. Venous thromboembolism following 672,495 primary total shoulder and elbow replacements: Meta-analyses of incidence, temporal trends and potential risk factors. Thromb Res. 2020 May;189:13-23. doi: 10.1016/j.thromres.2020.02.018. Epub 2020 Feb 20. PMID 32135385
- [Background] Mahabier KC, Den Hartog D, Theyskens N, Verhofstad MHJ, Van Lieshout EMM; HUMMER Trial Investigators. Reliability, validity, responsiveness, and minimal important change of the Disabilities of the Arm, Shoulder and Hand and Constant-Murley scores in patients with a humeral shaft fracture. J Shoulder Elbow Surg. 2017 Jan;26(1):e1-e12. doi: 10.1016/j.jse.2016.07.072. Epub 2016 Oct 10. PMID 27745806
- [Derived] Karimi D, Brorson S, Midtgaard KS, Fjalestad T, Paulsen A, Olerud P, Ekholm C, Wolf O, Viberg B; SHAFT Collaborators. Surgical versus non-surgical treatment of humeral SHAFT fractures compared by a patient-reported outcome: the Scandinavian Humeral diAphyseal Fracture Trial (SHAFT)-a study protocol for a pragmatic randomized controlled trial. Trials. 2022 Jun 2;23(1):453. doi: 10.1186/s13063-022-06317-6. PMID 35655280